CLINICAL TRIAL: NCT01394250
Title: Testing the Efficacy of a Vibrating, Cold Device for Pediatric IV Cannulation Pain Relief in the Emergency Department
Brief Title: Vibrating, Cold Device for Pediatric Intravenous (IV) Cannulation Pain Relief
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-007970
Record Dates: First submitted 2011-06-03; First posted 2011-07-14 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-07

CONDITIONS: Pain; Anxiety
Keywords: Pain; Anxiety; IV Cannulation; Topical Lidocaine; Buzzy; Face, Legs, Activity, Crying, Consolability (FLACC) scale; Faces Pain Scale Revised (FPS-R); Child Rating of Anxiety Scale
MeSH Terms: conditions — Pain; Anxiety Disorders; Facies; Motor Activity; Crying | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buzzy (Experimental): If randomized to Buzzy®, the nurse will demonstrate the cold pack and the device just prior to the IV cannulation procedure. The device will be applied with a Velcro strap 5 centimeters proximal to the site of IV cannulation; it will remain in place until the IV cannula is inserted and secured. All nurses that work during the study hours will be trained on the device prior to beginning the study. Training includes direct one-one training with the device including return demonstration.
  Interventions: Device: Buzzy
- Topical Lidocaine 4% Cream (Active Comparator): If randomized to topical lidocaine cream, subjects will have the cream placed on two or more potential IV sites as soon as possible after the consent procedure is complete. These subjects will undergo IV placement no less than 30 minutes after the cream is applied.
  Interventions: Drug: Topical Lidocaine 4% Cream

INTERVENTIONS:
Device: Buzzy — Cold, Vibrational Device
  Arms: Buzzy
Drug: Topical Lidocaine 4% Cream — Applied to anticipated IV site at least 30 minutes prior to cannulation.
  Other Names: AneCream™; Anestacon®; Dalcaine®; L-M-X™4; Xylocaine®
  Arms: Topical Lidocaine 4% Cream

SUMMARY:
The purpose of this study is to test the effectiveness of Buzzy®, a battery-powered reusable device that provides cold and vibration, in reducing the pain associated with intravenous (IV) cannulation. The investigators will investigate if Buzzy® is as effective as topical lidocaine cream in reducing the pain associated with IV cannulation.

DETAILED DESCRIPTION:
Intravenous (IV) cannulation is a significant source of pediatric pain and distress. Accumulating evidence has demonstrated that pain from IV cannulation is a significant source of pediatric pain and distress with effects far more reaching than the presenting event. When describing worse pain experiences in hospitalized children, IV cannulation pain was found to be second only to pain related to the subject's underlying disease. Practitioners recognize the need to mitigate or decrease pediatric IV cannulation pain and distress in emergency department patients, yet often do not provide the relief measures that are available. The use of topical lidocaine cream has some barriers, including the need to predict the need for the IV, the 30 minute administration time, difficulty in applying and maintaining the cream, the need for a physician's order and nursing to override in the Pyxis machine in order to obtain the medication in a timely manner.

Buzzy® provides a potential alternative to treating pediatric IV cannulation pain in the emergency department (ED), as cold and vibration are quick-acting options for pain relief. If Buzzy® is demonstrated to be as effective or more effective for reducing the pain of IV cannulation it would be an inexpensive and rapid way to provide pain control in accordance to the American Academy of Pediatrics (AAP) and American Pain Society recommendations. The device's actions are based on the Gate Control Theory, whereby cold and vibratory stimulation stimulate large fiber and inhibitory neurons to interrupt nociception. The benefits of Buzzy® include a low cost of $34.99 per reusable device, which could also provide a significant cost savings over the use of single tubes of topical lidocaine cream at a cost of $4.62-12.00 per tube with one or more tubes needed for each patient. Buzzy® does not require a medical order, but must be cleaned according to institution standards and is supplied with either a reusable cold pack or single use cold packs as desired. The commonly voiced concern related to the application of cold causing vasoconstriction has not been borne out in prior studies of Buzzy®.

Self-report of pain is the gold standard in evaluating pediatric pain. For this study we will use the Faces Pain Scale-Revised (FPS-R) for rating self-reported pain in children ages 4-18 years. The FPS-R has been validated and frequently used in pediatric pain studies. The FPS-R consists of 6 cartoon faces that range from a neutral expression ("no pain") to one of very much pain. Using the same faces, children will be asked how much the procedure "hurt" from "no hurt" to "very much hurt". Self-reporting of pain is the primary source of data and a secondary measure of data will be an observational pain scale, the face, legs, activity, cry, consolability (FLACC) scale. Because anxiety has proven to affect pain ratings, we will also evaluate anxiety using "Child Rating of Anxiety Scale", a visual semantic scale in the form of a thermometer for rating anxiety.

All subjects in this study will develop and implement a coping plan with a Child Life Specialist, including preparation, distraction, and deep breathing. This is standard of care in our ED and applied whenever possible for IV placement procedures. Child Life Specialists prepare subjects and families prior to medical procedures to decrease anxiety and increase understanding. Psychological preparation is aimed to increase a subject and family's control over a situation or procedure. While decreasing anxiety and increasing control, the child can move past the event with a sense of mastery and a low level of distress. Preparation close to the event is important for younger subjects, whereas preparation for older subjects is more beneficial when initiated earlier. The effectiveness of distraction in needle related procedures is well documented in the literature. Distraction involves a supportive care giver (if present) as well as a Certified Child Life Specialist; all attempts are made to focus of child away from the pain of the procedure and when possible the child is permitted to hold the objects and manipulate them prior to the procedure to enhance the utilization of a coping plan.

ELIGIBILITY:
Inclusion Criteria:

* Subject is aged 4 to 18 years of age
* Subjects will be having a peripheral IV line placed at the discretion of the treating physician for usual care of presenting complaints.
* Physician in charge of the subject is willing to wait the 30 minutes needed for the study preparation
* Subject/caregiver understands English
* Parent or legal guardian has signed Institutional Review Board (IRB) approved informed consent and subject (if age 7 years or older) has given assent

Exclusion Criteria:

* Subject is critically ill with a triage category of 1
* Subject has a condition that precludes the use of the self-report pain scale
* Subject has an abrasion, infection or break in skin in the area where Buzzy® would be placed
* Nerve damage is present in the extremity for planned IV placement

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 240 (Actual)
Dates: Start 2011-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Fein, MD, MPH, Principal Investigator — Children's Hospital of Philadelphia; Debra Potts, MSN, RN, Study Director — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Baxter AL, Leong T, Mathew B. External thermomechanical stimulation versus vapocoolant for adult venipuncture pain: pilot data on a novel device. Clin J Pain. 2009 Oct;25(8):705-10. doi: 10.1097/AJP.0b013e3181af1236. PMID 19920721
- [Background] Kennedy RM, Luhmann J, Zempsky WT. Clinical implications of unmanaged needle-insertion pain and distress in children. Pediatrics. 2008 Nov;122 Suppl 3:S130-3. doi: 10.1542/peds.2008-1055e. PMID 18978006
- [Background] American Academy of Pediatrics. Committee on Psychosocial Aspects of Child and Family Health; Task Force on Pain in Infants, Children, and Adolescents. The assessment and management of acute pain in infants, children, and adolescents. Pediatrics. 2001 Sep;108(3):793-7. doi: 10.1542/peds.108.3.793. PMID 11533354
- [Background] Cummings EA, Reid GJ, Finley AG, McGrath PJ, Ritchie JA. Prevalence and source of pain in pediatric inpatients. Pain. 1996 Nov;68(1):25-31. doi: 10.1016/S0304-3959(96)03163-6. PMID 9251995
- [Background] Rupp T, Delaney KA. Inadequate analgesia in emergency medicine. Ann Emerg Med. 2004 Apr;43(4):494-503. doi: 10.1016/j.annemergmed.2003.11.019. PMID 15039693
- [Background] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Background] Vanderah TW. Pathophysiology of pain. Med Clin North Am. 2007 Jan;91(1):1-12. doi: 10.1016/j.mcna.2006.10.006. PMID 17164100
- [Background] Hicks CL, von Baeyer CL, Spafford PA, van Korlaar I, Goodenough B. The Faces Pain Scale-Revised: toward a common metric in pediatric pain measurement. Pain. 2001 Aug;93(2):173-183. doi: 10.1016/S0304-3959(01)00314-1. PMID 11427329
- [Background] Kleiber C, McCarthy AM. Evaluating instruments for a study on children's responses to a painful procedure when parents are distraction coaches. J Pediatr Nurs. 2006 Apr;21(2):99-107. doi: 10.1016/j.pedn.2005.06.008. PMID 16545670
- [Background] Nilsson S, Finnstrom B, Kokinsky E. The FLACC behavioral scale for procedural pain assessment in children aged 5-16 years. Paediatr Anaesth. 2008 Aug;18(8):767-74. doi: 10.1111/j.1460-9592.2008.02655.x. PMID 18613934
- [Background] Cohen LL. Behavioral approaches to anxiety and pain management for pediatric venous access. Pediatrics. 2008 Nov;122 Suppl 3:S134-9. doi: 10.1542/peds.2008-1055f. PMID 18978007

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential subjects were identified in the Emergency Department (ED) from 2011-2014. When ED nurse anticipated intravenous (IV) placement, a member of the study team was contacted to screen for study eligibility.
Pre-assignment Details: A total of 315 subjets signed informed consent forms. Of these 47 subjects were excluded prior to initiation of study procedures. Reasons included parent/child withdrawal of consent, change in clinical treatment plan including the decision to not place an IV for clinical reasons (study exclusion).
Groups:
- Buzzy®: Buzzy® device was applied prior to intravenous cannulation.
- Topical Lidocaine 4% Cream: Topical Lidocaine 4% Cream was applied prior to intravenous cannulation.
Period: Randomization and IV Placement Attempt
Arm/Group | Buzzy® | Topical Lidocaine 4% Cream
Started | 134 | 134
Completed | 120 | 121
Not Completed | 14 | 13
Not completed — Unsuccessful IV Access on First Attempt | 14 | 13
Period: Successful IV Placement & Follow-Up
Arm/Group | Buzzy® | Topical Lidocaine 4% Cream
Started | 120 | 121
Completed | 114 | 110
Not Completed | 6 | 11
Not completed — Withdrawal by Subject | 6 | 11

BASELINE CHARACTERISTICS:
Population: Baseline analysis population includes all subjects who were randomized and whose first attempt at IV access was successful (i.e., subjects in the "Successful IV Placement & Follow-Up" group)
Groups:
- Total: Total of all reporting groups
Arm/Group | Buzzy® | Topical Lidocaine 4% Cream | Total
Number analyzed (Participants) | 114 | 110 | 224
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 114 | 110 | 224
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 52 | 105
  Male | 61 | 58 | 119
Region of Enrollment [Number; unit: participants]
  United States | 114 | 110 | 224

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Faces Pain Scale Revised (FPS-R) at 30 Minutes After IV Cannulation
Description: The Faces Pain Scale Revised (FPS-R) is numerical self-report measure of pain intensity developed for children to score the sensation of pain from 0-10. Pictures of 6 cartoon faces ranging from neutral expression of "no pain" (0) to "very much pain" (10).
Time Frame: Baseline and 30 minutes
Population: Analysis population includes only subjects whose first intravenous (IV) cannulation attempt was successful.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Buzzy® | Topical Lidocaine 4% Cream
Number analyzed (Participants) | 114 | 110
units on a scale | -3.544 [-4.179 to -2.909] | -3.436 [-4.083 to -2.790]

2. Secondary Outcome: Comparison of the Face, Legs, Activity, Cry, Consolability Scale (FLACC) Score Immediately After IV Cannulation Between Groups
Description: The Face, Legs, Activity, Cry, Consolability scale or FLACC scale is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2. The FLACC score was completed immediately after IV cannulation by a member of the clinical care team who was not part of the study. During initial trial design, the goal was to collect FLACC score pre and post cannulation; however, it was decided prior to enrollment that FLACC score would not be collected pre cannulation, only post.
Time Frame: Up to 5 minutes after IV Cannulation
Population: Analysis population includes only subjects whose first intravenous (IV) cannulation attempt was successful.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Buzzy® | Topical Lidocaine 4% Cream
Number analyzed (Participants) | 114 | 110
units on a scale | 0.667 [0.425 to 0.909] | 0.333 [0.084 to 0.582]

ADVERSE EVENTS:
Time Frame: 30 minutes
Arm/Group | Buzzy® | Topical Lidocaine 4% Cream
Serious Adverse Events (participants affected / at risk) | 0/134 | 0/134
Other Adverse Events (participants affected / at risk) | 0/134 | 0/134

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes